CLINICAL TRIAL: NCT02543671
Title: Investigation of Vitamin D3 Enriched, Reduced-fat Yellow Cheese Efficacy to Prevent Vitamin D Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: University College Cork (Other); FrieslandCampina (Industry)
Responsible Party: Principal Investigator, Yannis Manios, Associate Professor, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 613977
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Hypovitaminosis D; Deficiency of Micronutrients
Keywords: vitamin D status; 25-hydroxyvitamin D; cheese; Randomized controlled trial; postmenopausal women; enriched; vitamin D3
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- vitamin D3 enriched cheese (Active Comparator): vitamin D3 enriched, reduced-fat yellow cheese
  Interventions: Other: vitamin D3 enriched, reduced-fat yellow cheese
- plain cheese (Placebo Comparator): plain (non-fortified) reduced-fat yellow cheese
  Interventions: Other: plain (non-fortified) reduced-fat yellow cheese

INTERVENTIONS:
Other: vitamin D3 enriched, reduced-fat yellow cheese — 60 grams of vitamin D3 enriched, reduced-fat yellow cheese provide 5.7 micrograms of vitamin D per day for 8 weeks
  Arms: vitamin D3 enriched cheese
Other: plain (non-fortified) reduced-fat yellow cheese — 60 grams of plain (non-fortified), reduced-fat yellow cheese provide 0 micrograms of vitamin D per day for 8 weeks
  Arms: plain cheese

SUMMARY:
The primary aim of the current study was to investigate whether the consumption of vitamin D3 enriched, reduced-fat yellow cheese can counterbalance the expected decrease in serum 25-hydroxyvitamin D concentration during winter in postmenopausal women in Greece, and in what degree it can contribute as a potential food-based strategy for the prevention of vitamin D deficiency. A secondary aim was also to investigate any potential effect of the intervention in several quality of life (QoL) indices in the population of postmenopausal women under study.

DETAILED DESCRIPTION:
Vitamin D status in postmenopausal women is of interest because of the association of low vitamin D status with increased risk of osteoporosis and related fractures. In addition, since there is increasing evidence that the dietary supply is often insufficient to offset the seasonal deficit in sunlight during winter months, fortified food and supplements are becoming important sources of dietary vitamin D intake to achieve optimal vitamin D status, especially in this high risk population. Although most studies have examined the effectiveness of vitamin D enriched milk and yogurt, there have been limited studies also exploring the effectiveness of vitamin D enriched cheese in enhancing vitamin D status and preventing vitamin D deficiency. However, fortification of cheese with vitamin D has certain technological considerations, particularly for reduced-fat varieties considering that vitamin D is a fat soluble nutrient.

The primary aim of the current study was to investigate whether the consumption of vitamin D3 enriched, reduced-fat yellow cheese can counterbalance the expected decrease in serum 25-hydroxyvitamin D concentration during winter in postmenopausal women in Greece, and in what degree it can contribute as a potential food-based strategy for the prevention of vitamin D deficiency. A secondary aim was also to investigate any potential effect of the intervention in several quality of life (QoL) indices in the population of postmenopausal women under study. .

ELIGIBILITY:
Inclusion Criteria:

* subjects are eligible if they are 55-75 years of age
* being at menopause for more than 5 years
* they used to consume cheese daily
* those with a Body Mass Index (BMI) range 20-33kg/m2

Exclusion Criteria:

* having any disease/ pathology that interacts with vitamin D metabolism
* taking medications that interact with vitamin D metabolism or vitamin D supplements for medical reasons (e.g. osteoporosis)
* planned vacation to a sunny holiday destination during the intervention period
* having a cow's milk allergy
* having a drugs and/or alcohol abuse

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
serum 25-hydroxyvitamin D concentration | 8 weeks

SECONDARY OUTCOMES:
physical functioning scale, Short Form 36 health survey questionnaire (SF-36) | 8 weeks
  score range from 0 [worst disability related to physical functioning] to 100 [no disability related to physical functioning]
role limitations due to physical health scale, Short Form 36 health survey questionnaire (SF-36) | 8 weeks
  score range from 0 [worst disability related to limitations due to physical health] to 100 [no disability related to limitations due to physical health]
role limitations due to emotional problems scale, Short Form 36 health survey questionnaire (SF-36) | 8 weeks
  score range from 0 [worst disability related to limitations due to emotional problems] to 100 [no disability related to limitations due to emotional problems]
vitality scale, Short Form 36 health survey questionnaire (SF-36) | 8 weeks
  score range from 0 [worst disability related to vitality to 100 [no disability related to vitality]
emotional well-being scale, Short Form 36 health survey questionnaire (SF-36) | 8 weeks
  score range from 0 [worst disability related to emotional well-being to 100 [no disability related to emotional well-being]
social functioning scale, Short Form 36 health survey questionnaire (SF-36) | 8 weeks
  score range from 0 [worst disability related to social functioning to 100 [no disability related to social functioning]
bodily pain scale, Short Form 36 health survey questionnaire (SF-36) | 8 weeks
  score range from 0 [worst disability related to bodily pain] to 100 [no disability related to bodily pain]
general health scale, Short Form 36 health survey questionnaire (SF-36) | 8 weeks
  score range from 0 [worst general health] to 100 [best general health]

CONTACTS AND LOCATIONS:
Overall Officials: Yannis Manios, Associate Professor, Principal Investigator — Harokopio University, Athens
Locations (1):
- Harokopio University of Athens, Kallithea, Attica, Greece